CLINICAL TRIAL: NCT04653311
Title: A Multicenter, Controlled Study to Evaluate the Efficacy and Safety of an Endoscopic Sutured Gastroplasty (With Endomina Device) in Patients With Non Alcoholic Steatohepatitis (NASH) and Fibrosis.
Brief Title: Evaluation of an Endoscopic Sutured Gastroplasty in Patients With NonAlcoholic Steatohepatitis (NASH) and Fibrosis.
Acronym: ENDONASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Collaborators: Epidemiological and Clinical Research Information Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2019/400 / B406201941027
Record Dates: First submitted 2020-08-18; First posted 2020-12-04 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Arm 1: Endomina procedure + lifestyle intervention Arm 2: Lifestyle intervention
Masking Description: The primary outcome will be blindly assessed at one year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endomina procedure + lifestyle intervention (Experimental): The procedure will be performed under general anesthesia with tracheal intubation. Endomina will be introduced into the stomach over a guidewire and then fixed to the endoscope. This group will also receive the medical standard treatment defined as lifestyle intervention.
  Interventions: Device: Endomina®
- Lifestyle intervention (No Intervention): The group will receive the medical standard treatment defined as lifestyle therapy combining diet (mediterranean diet) with increased physical activity

INTERVENTIONS:
Device: Endomina® — Endoscopic sleeve gastroplasty (Endomina) at J0 with multidisciplinary follow-up for 1 year
  Arms: Endomina procedure + lifestyle intervention

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a spectrum of liver diseases characterized by liver steatosis which can, in a minority of patients, progress to nonalcoholic steatohepatitis (NASH), fibrosis, and ultimately hepatocellular carcinoma and liver failure. NASH is also recognized as an independent cardiovascular risk factor. Currently, weight loss is the only validated treatment for NASH and also positively affect all the features of metabolic syndrome. Considering the known positive metabolic effects of bariatric surgery, efforts have been exerted to develop minimally endoscopic procedures aiming to induce weight loss. Therefore, we would like to evaluate in patients with NASH disease and fibrosis, the impact of an endoscopic sutured gastroplasty (with Endomina® device) on:

* Mainly liver histological endpoints but also,
* Surrogate markers of hepatic inflammation and fibrosis and
* Surrogate markers of insulin resistance as well as fasting lipid and glycemic profiles.

DETAILED DESCRIPTION:
Background and Rationale: Nonalcoholic steatohepatitis (NASH) is a chronic and progressive disease which can evolve to advanced fibrosis, cirrhosis, liver failure or liver cancer and is associated to a higher risk of death related mainly to cardiovascular events. Weight loss affects positively histological and metabolic features of NASH. Similarly, bariatric surgery improves NASH and fibrosis in morbidly obese patients. New medical devices have been developed to perform endoscopic sutured gastroplasty (ESG) in obese patients. Those affected with coexisting NASH might constitute a good indication for such procedure.

Objective: To determine whether ESG improves liver histology, defined as resolution of NASH without worsening of fibrosis at 48 weeks (primary outcome) after ESG.

Design, setting and participants: The ENDONASH trial is an investigator-initiated, randomized, controlled, European multicenter study with centrally blinded assessment of the primary outcome. Biopsy proven NASH patients will be randomly assigned (1:1) to either ESG associated to lifestyle intervention (LSI) or LSI alone using a computer-generated, centrally administered allocation, stratified by diabetes status, gender and fibrosis stage. Main inclusion criteria are: biopsy-proven NASH (i.e. Nonalcoholic Fatty Liver Disease Score ≥4), fibrosis stage ≥1, BMI between 27-40, controlled type 2 diabetes.

Sample size calculation: The study is powered to establish a 50% response rate of NASH resolution without worsening of fibrosis in the ESG group and a 10% response rate in the control group (according to our previous study1 and a study2 which has evaluated the impact of weight loss on NASH). Accepting an alpha risk of 0.05 (bilateral), a beta risk of 0.2 and a loss rate of 20%, a sample size of 100 patients is needed to achieve statistical significance. Analysis will be carried out by intention-to-treat analysis, which includes all patients who will undergo end-of treatment liver biopsy.

Procedures: Eligible patients will be allocated to one arm of the study by means of an online platform (ViedocTM). Demographics, anthropometric measurements, medical history, blood samples and transient elastography will be performed at baseline and at different time points after the randomization during the 48 weeks of follow-up. Finally, all patients will undergo an end-of treatment liver biopsy 48 weeks after randomization.

Conclusion: The expected conclusion will allow to demonstrate if ESG, as an add on to LSI, may increases the number of patients with resolution of NASH without worsening of fibrosis at one year.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 27 to 40 kg/m².
* Histological confirmation of steatohepatitis on a diagnostic liver biopsy by central reading of the slides (biopsy obtained within 6 months prior to Screening or during the Screening Period) with at least 1 in each component of the NAS (steatosis scored 0-3, ballooning degeneration scored 0-2, and lobular inflammation scored 0-3).
* NAS ≥4.
* Fibrosis stage of 1 or greater and below 4, according to the NASH CRN fibrosis staging system.
* Patients in whom it is safe and practical to proceed with a liver biopsy (in accordance with the current guidelines), and who agree to have:

  1. 1 liver biopsy during the Screening Period for diagnostic purpose (if no historical biopsy within 6 months before screening is available)
  2. a final liver biopsy after 1 year of treatment for assessment of the treatment effects on NASH and fibrosis
* For patients with type 2 diabetes, glycemia must be controlled (HbA1c < 9.0%). If glycemia is controlled by antidiabetic drugs, change in anti-diabetic therapy must follow these requirements:

  1. No qualitative change 6 months prior to diagnostic liver biopsy up to Randomization (i.e., implementation of a new anti-diabetic therapy) for patients treated with metformin, gliptins, sulfonylureas, sodium/glucose cotransporter (SGLT) 2 inhibitors, glucagon-like peptide (GLP)-1 agonists or insulin. Dose changes of these medications are allowed in the 6 months prior to diagnostic liver biopsy, except for GLP-1 agonists, which must remain on stable dose in the 6 months prior to diagnostic liver biopsy.
  2. No implementation of GLP-1 agonists and SGLT2 inhibitors up to 1 year.
  3. Initiation of any other antidiabetic drugs is allowed after randomization based on treating physicians' judgment, except for glitazones which are prohibited 6 months prior to diagnostic liver biopsy until the end of treatment.
* Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: clinical assessment, endoscopy, radiography, as well as laboratory investigations.
* Must be able to understand and be willing to provide written informed consent.
* Must live within 75 km of the treatment site.
* In case of obesity, had followed the bariatric multidisciplinary workup (blood analyses, dietician,psychologist and doctor appointments).

Exclusion Criteria:

* Other well documented causes of chronic liver disease according to standard diagnostic procedures including, but not restricted to:

  1. Positive hepatitis B surface antigen (HBsAg)
  2. Positive HCV RNA, (tested for in case of known cured HCV infection, or positive HCV Ab at Screening)
  3. Suspicion of drug-induced liver disease
  4. Alcoholic liver disease
  5. Autoimmune hepatitis
  6. Wilson's disease
  7. Primary biliary cholangiopathy, primary sclerosing cholangitis
  8. Genetic homozygous hemochromatosis
  9. Presence of HCC
  10. History or planned liver transplant, or current MELD score >12.
  11. Alpha-1 antitrypsin deficiency.
* Current or recent history (< 5 years) of significant alcohol consumption. For men, significant consumption is defined as higher than 30g pure alcohol per day. For women, it is defined as higher than 20g pure alcohol per day.
* Compensated and decompensated cirrhosis (clinical and/or histological evidence of cirrhosis). Notably, NASH patients with fibrosis stage=4 according to the NASH CRN fibrosis staging system are excluded.
* Weight loss of more than 5 % within 6 months prior to randomization.
* Pregnant or breast feeding women or planning to become pregnant during the study period.
* Patients with a history of clinically significant acute cardiac event within 6 months prior to Screening such as: stroke, transient ischemic attack, or coronary heart disease (angina pectoris, myocardial infarction, revascularization procedures).
* Known chronic heart failure (Grade I to IV of New York Heart Association classification).
* Uncontrolled hypertension during the Screening Period despite optimal antihypertensive therapy.
* Fibrates are not permitted from 2 months before Randomization. Patients that used statins, ezetimibe, or fibrate lipid lowering drugs before Screening may participate if the dosage has been kept constant for at least 2 months prior to Screening.
* Patients with HbA1c >9.0%. If >9% at the first Screening Visit, the HbA1c measurement can be repeated at the latest 2 weeks prior to Randomization. A repeated abnormal HbA1c (HbA1c >9.0%) leads to exclusion.
* Patients receiving thiazolidinediones (glitazones [pioglitazone, rosiglitazone]), unless the drug was discontinued at least 6 months before the diagnostic liver biopsy.
* Patients receiving vitamin E, unless the drug was discontinued at least 6 months before the diagnostic liver biopsy.
* Currently taking drugs that can induce steatosis/steatohepatitis including, but not restricted to:corticosteroids (parenteral & oral chronic administration only), amiodarone (Cordarone), tamoxifen (Nolvadex), and methotrexate (Rheumatrex, Trexall), which are not permitted 30 days prior to Screening and up to end of treatment.
* Any medical conditions that may diminish life expectancy to less than 2 years including known cancers.
* Evidence of any other unstable or, untreated clinically significant immunological, endocrine, hematological, gastrointestinal, neurological, neoplastic, or psychiatric disease.
* Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain.
* Positive anti-human immunodeficiency virus (HIV) antibody.
* AST and/or ALT> 10x upper limit of normal (ULN).
* Conjugated bilirubin> 1.50 mg/dl due to altered hepatic function. Gilbert Disease patients are allowed into the study.
* INR>1.40.
* Platelet count < 100,000/mm3.
* Serum creatinine levels> 1.53 mg/dl in males and > 1.24 mg/dl in females.
* Significant renal disease, including nephritic syndrome, chronic kidney disease (defined as patients with markers of kidney damage or eGFR of less than 60 ml/min/1.73m2).
* Unexplained serum CPK> 3x the ULN. In case of explained elevated CPK>3x the ULN, the measurement can be repeated prior to randomization. In this case, retest should be performed within 1 to 2 weeks after initial test. A CPK rates>3x ULN leads to exclusion.
* Use of anticoagulation or P2Y12 inhibitors (clopidogrel, prasugrel, ticagrelor) therapy.
* Achalasia and any other esophageal motility disorders.
* Active severe esophagitis (grade C to D of Los Angeles Classification).
* Active gastric ulcer.
* Gastrointestinal stenosis or obstruction.
* Patients with contraindications to MRI imaging.
* Currently participating in another study.
* Previous bariatric surgery, or endoscopic obesity-related therapy such as endoscopic sleeve gastroplasty. Presence of intragastric balloon or retrieval within 6 months before signing informed consent.
* Immunosuppressive therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2023-06-23 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
Rate of disappearance of NASH without worsening of fibrosis grade | at 48 weeks
  Diagnosis of NASH at the liver biopsy

SECONDARY OUTCOMES:
Incidence of all Adverse Device Effects | at 48 weeks
  Safety will be characterized by the incidence of all Adverse Device Effects (ADEs), non-serious and serious, possibly related to or related to the procedure and/or device that are experienced by study participants.
Change in th SF-46 quality of life score | at 48 weeks
  SF-36 quality of life score
Change in the NAS (NAFLD activity score) score | at 48 weeks
  NAS is a histological score established on the liver biopsy. The NAS ranges form 0 to 8. 8 is associated with the highest severity.
Change in liver histologic characteristics, such as steatosis, ballooning, lobular inflammation, and portal chronic inflammation scores. | at 48 weeks
  Individual scores of the NAS score, the higher score (i.e. 8) means the worst condition.
Weight loss from randomization to the end of treatment | at 48 weeks
  weight
Change in elastography measured by vibration-controlled transient elastography | at 48 weeks
  Elastography is an indirect noninvasive measurement of liver fibrosis
Change in NAFLD fibrosis score | at 48 weeks
  NAFLD fibrosis score is a non invasive biomarker of liver fibrosis, a score superior to 0,675 means the worst condition
Change in Alanine Transaminase (ALT) | at 48 weeks
  ALT is a liver enzyme, used for the biological liver test evaluation.
Change in Aspartate Transaminase (AST) | at 48 weeks
  AST is a liver enzyme, used for the biological liver test evaluation.
Change in metabolic profile assessed by HOMA score | at 48 weeks
  HOMA is a score (scale) evaluating insulin resistance.
Change in Fasting glucose | at 48 weeks
  fasting glucose is a marker of diabetes and insulin resistance
Change in Glycated haemoglobin | at 48 weeks
  glycated haemoglobin is a surrogate marker for diabetes management and outcome.
Change in HDL cholesterol | at 48 weeks
  HDL cholesterol is a biomarker for lipid metabolism and cardiovascular risk
Change in serum triglycerides | at 48 weeks
  serum triglycerides is a biomarker for lipid metabolism and cardiovascular risk
Change in LDL cholesterol | at 48 weeks
  LDL cholesterol is a biomarker for lipid metabolism and cardiovascular risk
Change in total cholesterol. | at 48 weeks
  total cholesterol is a biomarker for lipid metabolism and cardiovascular risk
Correlation between mediterranean diet score and NAS score change | at 48 weeks
  Mediterranean diet assessment score evaluate the compliance to the mediterranean diet, the highest score (i.e.5) means the highest adherence

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Deviere, MD, phD, Principal Investigator — CUB Hôpital Erasme, Brussels, Belgium
Locations (1):
- CUB Hôpital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No